CLINICAL TRIAL: NCT02412579
Title: Circulating MicroRNA Isoforms as Biomarkers in Hepatocellular Carcinoma and Associated Liver Transplantation
Brief Title: Genetic Profiling of Liver Cancer in Patients Undergoing Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 014-121
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hepatocellular carcinoma tumor tissue Background liver tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hepatocellular Carcinoma with Cirrhosis: Subjects with hepatocellular carcinoma and cirrhosis.
  Interventions: Other: None - Standard of Care
- Cirrhosis without Hepatocellular Carcinoma: Subjects with only cirrhosis.
  Interventions: Other: None - Standard of Care

INTERVENTIONS:
Other: None - Standard of Care

SUMMARY:
The purpose of this study is to determine whether genetic markers unique to liver cancer are present and to assess usefulness as a diagnostic tool.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common form of liver cancer and a growing trend worldwide. Decision-making regarding treatment for patients is limited by the lack of clinically actionable biomarkers. This is pronounced in the case for determining and monitoring liver transplant recipients. In an effort to improve diagnosis, the use of circulating serum-based microRNA isoforms (isomiRs) can serve as non-invasive, screening biomarkers in HCC patients pre- and post-transplantation of the liver.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of HCC who are on the wait list for liver transplantation
* Patients with the diagnosis of HCC who have been admitted to hospital, scheduled to undergo liver transplantation within the following 24 hours.
* Age Range: 18 to 75 years old

Exclusion Criteria:

* Patients with metastatic HCC and patients with the diagnosis of HCC who are not on the wait list for liver transplantation.
* Patients older than 75 years old and younger than 18 years old.
* Patients who are unable to consent.
* Pregnant patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular Carcinoma Clinic Pre-Liver Transplant Clinic
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Using next-generation sequencing methods to detect isomiRs across different HCC cohorts at all stages undergoing liver transplantation. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kim, M.D., Principal Investigator — Annette C. & Harold C. Simmons Transplant Institute
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States